CLINICAL TRIAL: NCT01839643
Title: Phase 1 Study of Assessment of Local Absorption of a Non-steroidal Antiinflammatory Drug (NSAID), Inhibitor of Cyclooxygenase 2 (COX-2) Meloxicam, Through a Vaginal Ring and Its Effect on Ovarian Cycle in Fertile Women
Brief Title: Assessment of a Vaginal Ring With Meloxicam on Ovarian Cycle in Fertile Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Laboratorios Andromaco S.A. (Industry)
Collaborators: Instituto Chileno de Medicina Reproductiva (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: AVM-01001
Record Dates: First submitted 2013-03-18; First posted 2013-04-25 (Estimated); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Contraception; Bleeding Pattern
Keywords: pharmacokinetic
MeSH Terms: interventions — Meloxicam

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | US Export: No

ARMS (2):
- 2.4 g Meloxicam Vaginal Ring (Experimental): Continuous wearing during one menstrual cycle (6 participants)
  Interventions: Drug: Meloxicam 2.4 g
- 3.0 g Meloxicam Vaginal Ring (Experimental): Continuous wearing during one menstrual cycle (6 participants)
  Interventions: Drug: Meloxicam 3.0 g

INTERVENTIONS:
Drug: Meloxicam 2.4 g — 2.4 g in Vaginal Ring
  Arms: 2.4 g Meloxicam Vaginal Ring
Drug: Meloxicam 3.0 g — 3.0 g in Vaginal Ring
  Arms: 3.0 g Meloxicam Vaginal Ring

SUMMARY:
In this study, the investigators propose to assess if a non-hormonal agent is absorbed by a local route (vaginal) and to observe the effect on follicular development.

DETAILED DESCRIPTION:
Each volunteer will participate for 3 menstrual cycles, beginning with one menstrual control cycle without treatment, following by one menstrual cycle with meloxicam ring administration, and finishing with another control menstrual cycle.

Meloxicam will be administered in the second menstrual cycle via a vaginal ring in two doses of 2.4 g or 3.0 g/ring. The safety of the vaginal ring and the absorption of meloxicam will be assessed. Also the effect on follicular development and if it maintains ovarian cyclicity, as shown in a recent study with oral administration, will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Previous (or history of) proven fertility
* Regular menstrual cycle
* Surgically sterile
* Without breastfeeding
* Haemoglobin at least 11g/dL
* Willing to participate in the study

Exclusion Criteria:

* Allergy to meloxicam or other NSAID
* Allergy to silicone polymer
* Vaginal discharge non diagnosticated
* History of shock toxic syndrome
* History of : gastrointestinal, bleeding, renal, liver, heart, brain,clot, endocrine or pulmonary disorders

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2013-01-15 (Actual); Primary Completion 2013-05-07 (Actual); Study Completion 2013-06-06 (Actual)

PRIMARY OUTCOMES:
Number of participants with follicular rupture delay | Participants will be followed for the duration of one menstrual cycle, an expected average of 28 days
  Evaluate effective dose of maximum local safety that causes a greater proportion of follicular rupture delays when it is administered continuously, starting on the day 5 +/- 1 of the cycle until next menses.

SECONDARY OUTCOMES:
Pharmacokinetic of meloxicam via vaginal route: AUC | An expected average of 28 days
  The AUC of meloxicam serum levels
Bleeding patterns with meloxicam vaginal ring | one menstrual cycle
  Women will complete a menstrual diary during their participation to evaluate the effects of treatment on the menstrual pattern.
Pharmacokinetic of meloxicam via vaginal route: Tmax | An expected average of 28 days
  Tmax of meloxicam serum levels
Pharmacokinetic of meloxicam via vaginal route: Cmax | An expected average of 28 days
  Cmax of meloxicam serum levels

CONTACTS AND LOCATIONS:
Overall Officials: Grünenthal Study Director, Study Director — Grünenthal GmbH
Locations (1):
- Instituto Chileno de Medicina Reproductiva (ICMER), Santiago, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jesam C, Salvatierra AM, Schwartz JL, Croxatto HB. Suppression of follicular rupture with meloxicam, a cyclooxygenase-2 inhibitor: potential for emergency contraception. Hum Reprod. 2010 Feb;25(2):368-73. doi: 10.1093/humrep/dep392. Epub 2009 Nov 19. PMID 19933235
- See also: Link to clinical site — http://www.icmer.org